CLINICAL TRIAL: NCT04110041
Title: Assessing the Clinical & Neural Outcomes in Depressed Youth Randomized to One of Two Intensities of Aerobic Exercise
Brief Title: Effects of Aerobic Exercise Intensity on Clinical & Neural Outcomes in Depressed Youth
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Royal's Institute of Mental Health Research (Other)
Responsible Party: Principal Investigator, Dr. Natalia Jaworska, Director, Clinical Electrophysiology Laboratory, The Royal's Institute of Mental Health Research
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018025
Record Dates: First submitted 2019-09-23; First posted 2019-10-01 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Depression
Keywords: Transitional-aged youth; Exercise therapy; Neurocognition; fMRI; EEG
MeSH Terms: conditions — Depression | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moderate Intensity (Experimental): Aerobic exercise maintained for 30 minutes at 50-55% of each participant's individual heart rate reserve (HRRes).
  Interventions: Behavioral: Aerobic Exercise
- High Intensity (Experimental): Aerobic exercise maintained for 30 minutes at 80-85% of each participant's individual heart rate reserve (HRRes).
  Interventions: Behavioral: Aerobic Exercise

INTERVENTIONS:
Behavioral: Aerobic Exercise — Thrice-weekly aerobic exercise sessions lasting ~45 minutes, for 12 consecutive weeks.

SUMMARY:
This study will assess the effects of moderate vs. high intensity aerobic exercise, performed 3 times a week for 12 weeks under supervised conditions, on symptoms of depression, cognitive functioning and brain function in transitional aged youth (TAY: aged 16-24 years).

DETAILED DESCRIPTION:
Rationale: Major depressive disorder (MDD) is a debilitating disorder characterized by persistent negative mood and a broad range of cognitive, and functional impairments. MDD is estimated to affect 4.4% of the global population, or over 300 million individuals, representing the single largest contributor to non-fatal health loss worldwide. Current treatment options are associated with sub-optimal rates of remission, with only 30-35% of MDD sufferers attaining remission with antidepressant drug monotherapy. One group for whom treatment selection is a particular challenge is transitional aged youth (TAY), encompassing the late teenage years into the early twenties. Although MDD onset typically occurs during this period - as high as 8.2% in Canadian TAY - the psychiatric community has only recently begun to recognize TAY as a unique psychiatric cohort in need of directed treatment. For example, although the use selective serotonin reuptake inhibitors (SSRIs) is the first-line treatment for MDD in adults, their utility in TAY is hampered by the possibility of increased suicidal ideation within this cohort. The need for alternative and tailored treatment options for TAY with MDD is therefore of paramount importance. Aerobic exercise (AE) has recently been recognized as one such intervention, with some reports showing outcomes comparable to pharmacological and psychotherapeutic approaches in adult populations. Few studies however, have investigated to what extent these findings extend to TAY. Further, there is little consensus as to which intensity level, or "dose", of AE offers the most benefit, which neural features underlie the putative benefits of AE in depressed TAY, and the impact on both psychosocial and cognitive processes.

Objectives: The primary objectives of this study are: 1) to determine the effects of moderate vs. high intensity AE on clinically-rated and subjective symptoms of MDD in TAY; and 2) to examine the psychosocial, cognitive, and neuromodulatory effects of these interventions.

Methods: This two-arm, randomized trial will recruit 40 TAY (16-24 yrs) with MDD/persistent depressive disorder (PDD) into one of two AE intensity groups: medium or high. Intensity is defined as a percentage of heart rate reserve (HRR) achieved during exercise, as outlined in the American College of Sports Medicine (ACSM) guidelines (moderate: 50-55% of HRR; N=20; high: 80-85% HRR; N=20). All participants will undergo supervised and guided AE intervention sessions (~30min), three times per week, for twelve consecutive weeks. Pertinent clinical and psychosocial scores, as well as cardiac function (as assessed by maximal oxygen consumption [VO2max]), will be recorded pre-intervention (Week 0), mid-intervention (Week 6), and post-intervention (Week 12). Additionally, participants will undergo electroencephalographic (EEG) and functional magnetic resonance neuroimaging (fMRI) before and after the completion of AE intervention. Specifically, neural dynamics will be recorded at rest and during cognitive tasks engaging working memory (N-Back task) and response inhibition (Flanker task) - cognitive abilities, which have been shown to be impaired in MDD in TAY. Both clinical/psychosocial and neuroimaging outcomes will be compared using time as the within-group, and intervention type as between-group factors.

Hypotheses: The investigators expect a significant reduction in depression symptoms post (vs. pre) intervention and, based on preliminary evidence in adults, a greater reduction may emerge in those participating in the high (vs. moderate) intensity AE. Further, the investigators expect changes in fMRI profiles from pre- to post-intervention (showing normalization of brain activity and connectivity profiles); the same is true of EEG/event-related potential (ERP) features. They also expect a positive relation between VO2max and brain-based changes.

Significance: Findings from this project will help guide future large-scale investigations of AE as a potential treatment for TAY by clarifying the relation between changes to physical indices, depressive symptoms and neural profiles. Importantly, identifying the brain features modulated by AE will broaden our understanding of the neurobiological markers underlying depressive states, allowing for targeted therapeutic approaches and better outcomes for TAY suffering from MDD.

ELIGIBILITY:
Inclusion Criteria:

* Currently experiencing depression (MDD or PDD);
* Free of pharmacotherapy (ie. antidepressant medication) for >5 weeks;
* Not currently engaging in regular moderate or vigorous intensity exercise;
* Able to read/understand English;
* Body mass index [BMI] < 40;
* Medically cleared to engage in aerobic exercise.

Exclusion Criteria:

* Currently engaged in another exercise trial;
* Another Axis I/II DSM-5 disorder, apart from co-morbid anxiety disorder(s);
* Current or lifetime history of serious medical or neurological conditions;
* Currently taking psychoactive drugs (occasional use of anti-anxiety medication permitted);
* Regular user of nicotine products;
* Unstable medical conditions, especially those that prevent exercise;
* Exhibiting significant suicide risk;
* MRI contraindications;
* Currently pregnant or breastfeeding.

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-08-07 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Changes in clinician-rated depression-related symptoms | Baseline, Mid-Intervention (6 weeks), Post-Intervention (12 weeks)
  Changes in depressive symptoms as measured by the Hamilton Depression Rating Scale (HDRS) & Montgomery-Asberg Depression Rating Scale (MADRS).
Changes in self-reported depression-related symptoms | Baseline, Mid-Intervention (6 weeks), Post-Intervention (12 weeks), 3-month follow-up, 6-month follow-up
  Changes in depressive symptoms as measured by the Beck Depression Inventory (BDI; self-reported)
Feasibility of moderate & high intensity aerobic exercise as a treatment regimen. | Every 24 months from recruitment initiation until study completion
  Operationalized as: a) recruitment and randomization - the number of individuals who are successfully screened into the study, and the number of individuals randomized to each treatment following successful screening, respectively, over a 24 month period; and b) retention - the extent to which participants remain enrolled in the study, ie the number of participants who complete follow-up testing.
Adherence to moderate & high intensity exercise regimens as prescribed | Assessed per participant, through study completion
  The number of exercise session attended by each participant (out of the total 36 sessions prescribed).
Compliance to moderate & high intensity exercise regimens as prescribed | Assessed per participant, through study completion
  The percentage of time, per session, that a participant spends within his/her prescribed heart rate zone.

SECONDARY OUTCOMES:
Changes in electrocortical-indexed brain activity profiles | Baseline & Post-Intervention (12 weeks)
  Assessed via EEG during computerized tasks of attention/inhibition and working memory.
Changes to neuroimaging-indexed brain activity profiles | Baseline & Post-Intervention (12 weeks)
  Assessed via fMRI during computerized tasks of attention/inhibition and working memory.
Changes to self-esteem | Baseline, Mid-Intervention (6 weeks), Post-Intervention (12 weeks)
  Assessed with the Rosenberg Self-Esteem Scale, a 10-item self-report questionnaire.
Changes in self-mastery | Baseline, Mid-Intervention (6 weeks), Post-Intervention (12 weeks)
  Assessed with Perlin/Schooler's Mastery Scale a 7-item self-report questionnaire.
Changes in daily functioning | Baseline, Mid-Intervention (6 weeks), Post-Intervention (12 weeks)
  Assessed via the Columbia Impairment Scale, a 13-item self-report questionnaire.
Changes in cognitive function | Baseline, Mid-Intervention (6 weeks), Post-Intervention (12 weeks)
  Assessed via the NIH Cognitive Toolbox; a cognitive battery consisting of 7 distinct computerized tasks assessing multiple cognitive constructs. Performance on each task is combined to produce a composite score.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Ottawa Institute of Mental Health Research, Ottawa, Ontario, Canada